CLINICAL TRIAL: NCT01264757
Title: Steps Toward Adapting Physical Activity Guidelines for the Lower Mississippi Delta Population
Acronym: STEPS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Peter T. Katzmarzyk, Associate Executive Director for Population and Public Health, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 29034
Record Dates: First submitted 2010-12-03; First posted 2010-12-22 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Physical Inactivity
Keywords: pedometer; accelerometer; moderate-to-vigorous physical activity; adult; randomized trial
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education (Active Comparator): Educational brochure about physical activity provided.
  Interventions: Behavioral: Physical Activity Educational Materials
- Pedometer (Experimental): A pedometer was provided in addition to educational materials.
  Interventions: Behavioral: Pedometer

INTERVENTIONS:
Behavioral: Physical Activity Educational Materials — A brochure was provided to participants about the health benefits of physical activity and physical activity recommendations
  Arms: Education
Behavioral: Pedometer — A pedometer was provided to participants in addition to educational materials about the health benefits of physical activity.
  Arms: Pedometer

SUMMARY:
This feasibility study specifically addresses the issue of adapting US dietary guidelines physical activity recommendations to the population of the Lower Mississippi Delta. The hypothesis is that including a pedometer as a self-monitoring tool as part of adapted physical activity guidelines will result in greater immediate increases in physical activity (as monitored by an accelerometer) than an education program alone.

DETAILED DESCRIPTION:
The purpose of this study was to determine if a short-term pedometer-based intervention results in immediate increases in time spent in moderate-to-vigorous physical activity (MVPA) compared to a minimal educational intervention.A sample of 43 overweight adults 35 to 64 years of age participated in a one week pedometer-based feasibility trial monitored by accelerometry. Participants were randomized into a one-week education-only group or a group that also wore a pedometer. Accelerometer-measured MVPA was measured over 7 days at baseline and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* 35 to 64 years of age
* body mass index (BMI) between 25 and 34.9 kg/m2
* being able to walk without limitation

Exclusion Criteria:

* cardiovascular, respiratory, gastrointestinal, neuromuscular, neurological, or psychiatric problems; musculoskeletal problems interfering with exercise
* immunodeficiency problems
* malignancies in the last 5 years
* any other medical condition or life threatening disease that could be aggravated by exercise

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Minutes spent in moderate-to-vigorous physical activity (MVPA) | The primary outcome is measured at baseline and after a 7-day intervention period (1 week)
  A GT3X accelerometer is used to monitor each participants physical activity levels for seven consecutive days at baseline and again following a 7-day intervention period. The amount of time per day spent above a threshold of 2200 accelerometer counts/min is averaged over at least three days as the measure of MVPA.

CONTACTS AND LOCATIONS:
Overall Officials: Peter T Katzmarzyk, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katzmarzyk PT, Champagne CM, Tudor-Locke C, Broyles ST, Harsha D, Kennedy BM, Johnson WD. A short-term physical activity randomized trial in the Lower Mississippi Delta. PLoS One. 2011;6(10):e26667. doi: 10.1371/journal.pone.0026667. Epub 2011 Oct 25. PMID 22046325
- [Result] Harrington DM, Tudor-Locke C, Champagne CM, Broyles ST, Harsha DW, Kennedy BM, Johnson WD, Allen R, Katzmarzyk PT. Step-based translation of physical activity guidelines in the Lower Mississippi Delta. Appl Physiol Nutr Metab. 2011 Aug;36(4):583-5. doi: 10.1139/h11-053. Epub 2011 Aug 19. PMID 21854159